CLINICAL TRIAL: NCT05657899
Title: The With Or Without Olecranon K-wire (WOW OK) Trial of Tension Band Wire Fixation Versus Cerclage Fixation Without K-wires in Displaced Stable Olecranon Fractures
Brief Title: The With Or Without Olecranon K-wires Trial
Acronym: WOW-OK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DSF-220510-2038
Record Dates: First submitted 2022-11-16; First posted 2022-12-20 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Olecranon Fracture
Keywords: Tension Band Wiring; Cerclage; Surgery; Elbow injuries; Forearm injuries; Ulna fractures; Patient reported outcome measures
MeSH Terms: conditions — Olecranon Fracture; Elbow Injuries; Forearm Injuries; Ulna Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessor of all outcome measures except assessment of a postoperative radiograph will be masked. When the radiograph is viewed the operative method will be apparent, but this assessor is not the same as for the other outcome measures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cerclage (Active Comparator): Intervention by cerclage fixation.
  Interventions: Procedure: Cerclage fixation
- Tension Band Wiring (Active Comparator): Intervention by tension band wiring
  Interventions: Procedure: Tension band wiring

INTERVENTIONS:
Procedure: Cerclage fixation — The intervention is by surgical open reduction and internal fixation of the fracture using two 1.0mm cerclage.
  Arms: Cerclage
Procedure: Tension band wiring — The intervention is by surgical open reduction and internal fixation of the fracture using a 1.0mm cerclage and two 1.6 mm k-wires as described in AO-guidelines.
  Arms: Tension Band Wiring

SUMMARY:
Fractures of the elbow tip (olecranon) that leave the elbow joint stable but where the fracture ends are separated (Mayo type 2a and 2b) can be treated with pins and a metal wire (tension band wiring, TBW) or metal wiring alone (cerclage fixation, CF ). Previous studies have reported high re-operation and complication rates following TBW. The current study's hypothesis, based on two retrospective studies, is that CF of these fractures yield lower re-operation rates compared with TBW. The investigators also hypothesize that the overall complication rate will be lower following CF. The aim is to investigate this hypothesis in a randomized controlled trial. Patients that are 18 years or older with Mayo type 2a and 2b olecranon fractures at Skåne University hospital will be invited to the study. Participation is voluntary. Patients who accept participation will be randomly assigned to surgery by either TBW or cerclage fixation. Two hundred participants will be followed by physiotherapists for 36 months post-surgery assessing re-operations, complications, patient reported outcome, and elbow function.

DETAILED DESCRIPTION:
The complete study protocol including a detailed description of the trial will be published in a journal before the start of the trial.

Olecranon fractures account for approximately 20% of all proximal fractures of the forearm. Stable, undisplaced fractures (Mayo type 1a and 1b) are routinely treated non-operatively, while displaced and unstable fractures (Mayo type 3a and 3b) are typically operated with plate fixation. Stable, displaced fractures (Mayo type 2a and 2b) are often treated with tension band wiring (TBW) or plate fixation. TBW is associated with soft tissue irritation and high re-operation rates with hardware removal, ranging from 25% to 84% in the literature. Plate fixation was associated with fewer re-operations compared with TBW in a randomized controlled trial, but complications following plate fixation were more severe. A Cochrane review from 2014 did not find any significant support favouring either of the two methods. Non-operative treatment of Mayo type 2a and 2b fractures can yield acceptable results in elderly patients, but is not routinely used in younger individuals with higher functional demands. Two previous retrospective studies from 2002 and 2021 reported that Mayo 2a and 2b fractures can be operated with cerclage fixation alone yielding half the re-operation rates when compared to TBW. As of April 2022 there are two studies (one active (NCT03280602) and one completed (NCT01391936)) comparing TBW vs plate fixation, three studies (two active (NCT04670900 and NCT04401462) and one terminated (NCT01397643)) comparing non-operative vs operative treatment in elderly and one active study (NCT04189185) comparing TBW vs suture fixation registered on this site. The hypothesis of the current study is that the re-operation rate and the complication rate will be lower following CF compared with TBW while yielding equal results in other outcome measures. The aim is to to investigate this in a prospective randomized clinical trial.

Methodology:

All patients presenting at Skåne University Hospital in Malmö and Lund, Sweden, with olecranon fractures of Mayo type 2a and 2b will be invited to participate in the study if they do not meet any exclusion criteria. Potential subjects will be asked to sign a consent form after receiving written and oral information about the trial. Subjects will be randomized 1:1 to surgery with TBW or cerclage. 200 subjects will be recruited based on sample size calculations derived from the re-operation frequency in a previous study (PMID: 34236459)

Baseline descriptive data will be collected at inclusion or in the peri-operative period. Operation time, intra-operative effective radiation dose and radiation time will be recorded. Subjects will be invited to follow-up to a physiotherapist at 2 weeks, 6 weeks, 3 months, 12 months and 36 months after the operation assessing re-operations, complications, post-operative antibiotics, range of elbow motion, grip strength, the Quick Disabilities of the Arm, Shoulder and Hand score (Quick-DASH, references PMID: 8773720 and 6709254), overall patient satisfaction, pain, return to work and secondary dislocation. The Short Musculoskeletal Function Assessment (SMFA, references PMID: 27994082 and 14763711) score will be assessed 12 months post-operatively. The physiotherapist will be masked to the treatment method. At 6 months one radiograph will be collected for assessment of non-union.

The primary outcome measure will be re-operations. Secondary outcome measures will be patient reported outcome measures and complications. Tertiary outcome measures are post-operative range of motion and grip strength, secondary dislocation rate, time to return to work after surgery, operation time, effective intra-operative radiation dose and radiation time. The hypothesis of the current study is that cerclage fixation will yield less re-operations, less overall complications and less severe complications while other outcome measures will be equal.

ELIGIBILITY:
Inclusion Criteria:

* Sustained Olecranon type fracture of Mayo 2a or 2b
* Seeking healthcare in at the Skåne University Hospital in Lund and Malmö, Sweden.

Exclusion Criteria:

* Subjects unable to participate in follow up (for example subjects with active substance abuse, dementia, inability to communicate or understand the questionnaires or subjects living in other administrative healthcare regions).
* Subjects unable to give informed written consent.
* Subject where non operative treatment is indicated due to frailty or severe ongoing disease.
* Fracture not operated within 14 days from the date the fracture was sustained.
* Subjects with severe open fractures of Gustilo-Anderson class III
* Subject with pathological fractures from metastatic disease.
* Subject with simultaneous or previous severe injury to the same arm are excluded for patient reported outcome measures but included for all other outcomes.
* Subjects with previously severe injuries to the same arm will be excludes for PROM analyses but included for reoperation and complication analyses.
* Subjects operated by an orthopedic trauma surgeons that did not attended our education on the study and the interventions, unless surgery is supervised by an orthopedic surgeon that has attended the education the subject will not be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2029-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Re-operation rate 1.5 months. | Recorded at 1.5 months after intervention.
  Total re-operation rate of the operated elbow regardless of cause.
Re-operation rate 3 months. | Recorded at 3 months after intervention.
  Total re-operation rate of the operated elbow regardless of cause.
Re-operation rate 12 months. | Recorded at 12 months after intervention.
  Total re-operation rate of the operated elbow regardless of cause.
Re-operation rate 36 months. | Recorded at 36 months after intervention.
  Total re-operation rate of the operated elbow regardless of cause.

SECONDARY OUTCOMES:
Complication rate 1.5 months. | Recorded at 1.5 months after intervention.
  Total complication rate.
Complication rate 3 months. | Recorded at 3 months after intervention.
  Total complication rate.
Complication rate 12 months. | Recorded at 12 months after intervention.
  Total complication rate.
Complication rate 36 months. | Recorded at 36 months after intervention.
  Total complication rate.
Complication severity 1.5 months. | Recorded at 1.5 months after intervention.
  Complication severity classified with the Clavien-Dindo Classification.
Complication severity 3 months. | Recorded at 3 months after intervention.
  Complication severity classified with the Clavien-Dindo Classification.
Complication severity 12 months. | Recorded at 12 months after intervention.
  Complication severity classified with the Clavien-Dindo Classification.
Complication severity 36 months. | Recorded at 36 months after intervention.
  Complication severity classified with the Clavien-Dindo Classification.
Quick-DASH 1.5 months. | 1.5 months after intervention.
  Quick-DASH questionnaire assessed by subjects. See references PMID: 8773720 and 6709254.
Quick-DASH 3 months. | 3 months after intervention.
  Quick-DASH questionnaire assessed by subjects. See references PMID: 8773720 and 6709254.
Quick-DASH 12 months. | 12 months after intervention.
  Quick-DASH questionnaire assessed by subjects. See references PMID: 8773720 and 6709254.
Quick-DASH 36 months. | 36 months after intervention.
  Quick-DASH questionnaire assessed by subjects. See references PMID: 8773720 and 6709254.
SMFA 12 months | 12 months after intervention.
  SMFA-questionnaire assessed by subjects. See reference PMID: 27994082 and 14763711
Pain level 1.5 months. | Recorded at 1.5 months after intervention
  Subjective pain level in motion and at rest. Measured with a visual analog scale.
Pain level 3 months. | Recorded at 3 months after intervention.
  Subjective pain level in motion and at rest. Measured with a visual analog scale.
Pain level 12 months, | Recorded at 12 months after intervention.
  Subjective pain level in motion and at rest. Measured with a visual analog scale.
Pain level 36 months. | Recorded at 36 months after intervention.
  Subjective pain level in motion and at rest. Measured with a visual analog scale.
Overall satisfaction 1.5 months. | Recorded at 1.5 months after intervention.
  Subjective overall satisfaction level. Measured with a visual analog scale.
Overall satisfaction 3 months. | Recorded at 3 months after intervention.
  Subjective overall satisfaction level. Measured with a visual analog scale.
Overall satisfaction 12 months. | Recorded at 12 months after intervention.
  Subjective overall satisfaction level. Measured with a visual analog scale.
Overall satisfaction 36 months. | Recorded at 36 months after intervention.
  Subjective overall satisfaction level. Measured with a visual analog scale.

OTHER OUTCOMES:
Grip strength 0.5 months. | Recorded at 0.5 months after intervention.
  Grips strength will be evaluated using a JAMAR dynamometer as detailed in the Swedish National Quality Register for Hand Surgery (HAKIR)
Grip strength 1.5 months. | Recorded at 1.5 months after intervention.
  Grips strength will be evaluated using a JAMAR dynamometer as detailed in the Swedish National Quality Register for Hand Surgery (HAKIR)
Grip strength 3 months. | Recorded at 3 months after intervention.
  Grips strength will be evaluated using a JAMAR dynamometer as detailed in the Swedish National Quality Register for Hand Surgery (HAKIR)
Grip strength 12 months. | Recorded at 12 months after intervention.
  Grips strength will be evaluated using a JAMAR dynamometer as detailed in the Swedish National Quality Register for Hand Surgery (HAKIR)
Grip strength 36 months. | Recorded at 36 months after intervention.
  Grips strength will be evaluated using a JAMAR dynamometer as detailed in the Swedish National Quality Register for Hand Surgery (HAKIR)
Range of motion 0.5 months. | Recorded at 0.5 months after intervention.
  Active extension, flexion, pronation and supination will be evaluated using a goniometer following the Swedish National Quality Register for Hand Surgery (HAKIR) guidelines.
Range of motion 1.5 months. | Recorded at 1.5 months after intervention.
  Active extension, flexion, pronation and supination will be evaluated using a goniometer following the Swedish National Quality Register for Hand Surgery (HAKIR) guidelines.
Range of motion 3 months. | Recorded at 3 months after intervention.
  Active extension, flexion, pronation and supination will be evaluated using a goniometer following the Swedish National Quality Register for Hand Surgery (HAKIR) guidelines.
Range of motion 12 months. | Recorded at 12 months after intervention.
  Active extension, flexion, pronation and supination will be evaluated using a goniometer following the Swedish National Quality Register for Hand Surgery (HAKIR) guidelines.
Range of motion 36 months. | Recorded at 36 months after intervention.
  Active extension, flexion, pronation and supination will be evaluated using a goniometer following the Swedish National Quality Register for Hand Surgery (HAKIR) guidelines.
Time to return to work 1.5 months. | Recorded at 1.5 months after intervention.
  Time to return to work in days will be evaluated for all working subjects.
Time to return to work 3 months. | Recorded at 3 months after intervention.
  Time to return to work in days will be evaluated for all working subjects.
Time to return to work 12 months. | Recorded at 12 months after intervention.
  Time to return to work in days will be evaluated for all working subjects.
Time to return to work 36 months. | Recorded at 36 months after intervention.
  Time to return to work in days will be evaluated for all working subjects.
Secondary dislocation rate. | 6 months after intervention.
  Secondary dislocation rate will be assessed with a one lateral view radiograph of the operated elbow.
Intra-operative fluoroscopy radiation level. | Peri-operative.
  Intra-operative fluoroscopy radiation DAP will be recorded at the time of surgery from the fluoroscopy machine used.
Intra-operative fluoroscopy time. | Peri-operative.
  Intra-operative fluoroscopy time will be recorded at the time of surgery from the fluoroscopy machine used.
Antibiotic treatment 1.5. | Recorded at 1.5 months after intervention.
  Any unplanned prescription of antibiotics after the intervention related to the injury.
Antibiotic treatment 3. | Recorded at 3 months after intervention.
  Any unplanned prescription of antibiotics after the intervention related to the injury.
Antibiotic treatment 12. | Recorded at 12 months after intervention.
  Any unplanned prescription of antibiotics after the intervention related to the injury.
Antibiotic treatment 36. | Recorded at 36 months after intervention.
  Any unplanned prescription of antibiotics after the intervention related to the injury.
Surgical time. | Peri-operative.
  Time from incision to completed wound closure will be recorded during surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Wenger, MD, PhD, Principal Investigator — Department of Orthopedics, Skåne University Hospital and Lund University
Locations (2):
- Sweden (2):
  - Dept. of Orthopaedics, Lund, Skåne County
  - Dept. of Orthopaedics, Malmo, Skåne County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wenger D, Cornefjord G, Rogmark C. Cerclage fixation without K-wires is associated with fewer complications and reoperations compared with tension band wiring in stable displaced olecranon fractures in elderly patients. Arch Orthop Trauma Surg. 2022 Oct;142(10):2669-2676. doi: 10.1007/s00402-021-04027-3. Epub 2021 Jul 8. PMID 34236459
- [Background] Hudak PL, Amadio PC, Bombardier C. Development of an upper extremity outcome measure: the DASH (disabilities of the arm, shoulder and hand) [corrected]. The Upper Extremity Collaborative Group (UECG). Am J Ind Med. 1996 Jun;29(6):602-8. doi: 10.1002/(SICI)1097-0274(199606)29:63.0.CO;2-L. PMID 8773720
- [Background] Gries MW. Safety professional's role as health educator expanding. Occup Health Saf. 1984 Feb:42-3. No abstract available. PMID 6709254
- [Background] Williams N. The Short Musculoskeletal Function Assessment (SMFA) questionnaire. Occup Med (Lond). 2016 Dec;66(9):757. doi: 10.1093/occmed/kqw140. No abstract available. PMID 27994082
- [Background] Ponzer S, Skoog A, Bergstrom G. The Short Musculoskeletal Function Assessment Questionnaire (SMFA): cross-cultural adaptation, validity, reliability and responsiveness of the Swedish SMFA (SMFA-Swe). Acta Orthop Scand. 2003 Dec;74(6):756-63. doi: 10.1080/00016470310018324. PMID 14763711
- [Derived] Cornefjord G, Kostogiannis I, Rogmark C, Jerrhag D, Wenger D. The With Or Without Olecranon K-wire (WOW OK) Trial of tension band wire fixation versus cerclage fixation without K-wires in displaced stable olecranon fractures: study protocol for a randomized controlled trial. Trials. 2023 Aug 29;24(1):559. doi: 10.1186/s13063-023-07566-9. PMID 37641082